CLINICAL TRIAL: NCT02556125
Title: Intramuscular Pacing to Enhance Voluntary Diaphragm Activation
Brief Title: Diaphragm Pacing After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Brooks Rehabilitation (Other); The Craig H. Neilsen Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500402
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Injuries, Spinal Cord
Keywords: SCI; Respiratory impairment; Diaphragm pacing; Diaphragm stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical SCI: Participants with acute, traumatic cervical spinal cord injuries (C-SCIs), classified according to the American Spinal Injury Association (ASIA) Impairment Scale (AIS) as A-C (complete SCI (A); motor complete SCI (B); motor incomplete with minimal motor function (C)), affecting C1-C6 spinal cord segments, and who have been scheduled to undergo implantation of a diaphragm pacer, or who have recently received (in past 5-days) implantation of intramuscular diaphragm pacing electrodes due to severe respiratory impairments and dependence on mechanical ventilation.
  Interventions: Device: Diaphragm pacing

INTERVENTIONS:
Device: Diaphragm pacing — Intramuscular diaphragm implantation is achieved by a laparoscopic approach whereby phrenic motor points on the diaphragm are mapped to optimize electrode placement. The electrodes are threaded into the diaphragm muscle and wire leads are externalized and attached to a stimulation controller.

SUMMARY:
Respiratory dysfunction is the leading cause of death in individuals with spinal cord injuries (SCIs). Nearly one quarter of all SCI cases involve injury to the upper spinal cord segments which impairs neural activation of the diaphragm muscle and compromises breathing. Although mechanical ventilation can be life-saving after cervical SCI (C-SCI), it also triggers rapid and profound diaphragm muscle atrophy, thereby complicating (or even preventing) ventilator weaning. Intramuscular diaphragm stimulation, or diaphragm pacing, was developed to replace long-term ventilator support, and is now used acutely post C-SCI (<4 months following injury) to promote ventilator weaning. The impact of diaphragm pacing on respiratory function and diaphragm muscle activation has not been formally evaluated. This is an essential step in determining the efficacy of intramuscular diaphragm stimulation and its effects on respiratory function after SCI. Accordingly, this research study will evaluate the effects of intramuscular diaphragm stimulation and test the hypothesis that diaphragm pacing enhances neuromuscular diaphragm activation and respiratory function in adults with cervical SCIs. The investigators will test the hypothesis by evaluating the effects of diaphragm pacing on neuromuscular activation of the diaphragm by directly recording electromyogram (EMG) activity from the intramuscular pacing electrodes. Recording from these surgically-implanted electrodes allows direct comparisons of EMG activity across time, minimizing methodological limitations inherent with surface or percutaneous EMG recordings. This approach, in association with respiratory assessments, will be used to investigate the impact of diaphragm pacing in adults with intramuscular diaphragm pacing electrodes following acute, traumatic C-SCIs.

DETAILED DESCRIPTION:
Subject recruitment. Patients with acute, traumatic C-SCIs, scheduled to receive intramuscular diaphragm pacing OR who have recently received a diaphragm pacer (within past 5-days) will be recruited from two Level-1 trauma hospitals serving North Florida - UF Health Shands Hospitals in Gainesville and Jacksonville, Florida.

Enrollment. Patients with acute, traumatic C-SCIs (AIS A-C, affecting C1-C6 segments) who are scheduled to undergo or who have recently received implantation of diaphragm pacing electrodes (within recent 5-days) will be identified by the investigators.

After obtaining informed consent for participation in the study, members of the study team will review the participant's medical records to obtain study-related data and verify that the participant meets the study criteria. Clinical tests of sensory and motor function also may be conducted to verify the participant's SCI classification and extent of SCI. The tests of sensory and motor function are part of the American Spinal Injury Association (ASIA) Impairment Scale and the International Standards for Neurological Classification of Spinal Cord Injury. These clinical assessments are part of standard clinical care and include tests of sensation (dermatomes) and muscle strength via manual muscle testing (myotomes). These tests are done to clinically determine which segmental levels of the spinal cord demonstrate normal or impaired function. These tests also aid in determining if the SCI is clinically complete or incomplete. Determination of complete versus incomplete is based on the sensory and motor function in the lowest sacral segments which control sensation and motor function at the anal sphincter. Respiratory function will be assessed by measurement of maximal expiratory pressures and standard spirometry (tidal breathing, maximal voluntary ventilation and flow-volume curves).

Following enrollment and implantation of diaphragm pacing electrodes, individuals will be assessed at regular intervals. Assessments will include: a.) clinical ASIA neurologic examination of sensory and motor function (as described above) b.) recording of intramuscular diaphragm EMGs c.) measurement of diaphragm muscle strength via standard clinical assessment of maximal inspiratory pressures and d.) standard clinical measures of respiratory function.

Up to 5 assessments will be conducted in the acute hospital setting; up to 5 assessments during inpatient rehabilitation (Brooks Rehabilitation); up to 4 assessments will be conducted after discharge to the home setting.

ASSESSMENT OVERVIEW: The examination will allow investigators to characterize longitudinal changes in segmental sensory and motor function. Diaphragm electromyogram (EMG) will be recorded from the intramuscular diaphragm pacing electrodes and respiratory function will be assessed during non-stimulated respiration (diaphragm pacing unit turned off). Diaphragm EMGs will be recorded from the intramuscular pacing electrodes with a custom connector that attaches to the external pacing electrode wires and interfaces with an EMG acquisition system. Concurrent with EMG recordings, each assessment will include tests of maximal inspiratory pressures to assess diaphragm muscle strength.

Assessment of the neuromuscular activation of the diaphragm will be performed. Neuromuscular activation of the diaphragm will be assessed by recording diaphragm EMGs from the surgically-implanted intramuscular stimulating electrodes. This approach will allow for comparisons of EMG recordings across time and reduces the methodological limitations associated with surface or percutaneous EMG approaches. EMGs will be recorded during non-stimulated respiration (diaphragm pacer turned off) and simultaneously with assessments of respiratory function. These assessments may include maximal inspiratory pressures; sniff nasal inspiratory pressure, maximal expiratory pressure, assessments of resting tidal breathing, inspiration to total lung capacity, maximal voluntary ventilation and measurement of flow volumes using standard spirometry.

During the assessments, photographs and/or video recordings may be obtained. These recordings will be done with the participant's knowledge and consent for the type of recording being obtained. Photographs and video recordings will be used to communicate study procedures with the study team and to monitor the assessment process. Video and photographic data will be used to assess how individuals with SCIs perform and respond to the testing and to communicate the study procedures. Video and photographic information will be used in a manner based on the level of consent obtained from each participant.

Primary outcomes to characterize neuromuscular activation of the diaphragm and assess changes in diaphragm activation associated with intramuscular diaphragm stimulation will include: amplitude and timing characteristics (raw, filtered EMGs and normalized); neural respiratory drive to evaluate diaphragm muscle activation during tidal breathing relative to activation capacity during maximal inspiratory maneuvers; and time-frequency characteristics of the diaphragm EMGs (wavelet analysis).

ELIGIBILITY:
Inclusion Criteria:

* Acute, traumatic cervical spinal cord injuries (C-SCIs), classified according to the American Spinal Injury Association (ASIA) Impairment Scale (AIS) as A-C (complete SCI (A); motor complete SCI (B); motor incomplete with minimal motor function (C)), affecting C1-C6 spinal cord segments
* Scheduled to undergo implantation of a diaphragm pacer, or who have recently received (in past 5-days) implantation of intramuscular diaphragm pacing electrodes due to severe respiratory impairments and dependence on mechanical ventilation.

Exclusion Criteria:

* Progressive neuromuscular diseases such as multiple sclerosis and myasthenia gravis
* History of neurologic injuries such as stroke or prior SCI
* Chest wall injuries or deformities likely to influence breathing
* Pulmonary infection
* Pregnancy
* Cognitive impairments limiting study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty adults will be recruited from an acute care hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Electromyogram (EMG) will be used to assess the neuromuscular activation of the diaphragm | Change in baseline to months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  Neuromuscular activation of the diaphragm will be assessed by recording diaphragm EMGs from the surgically-implanted intramuscular stimulating electrodes. This approach will allow for comparisons of EMG recordings across time. EMGs will be recorded during non-stimulated respiration (diaphragm pacer turned off) and simultaneously with assessments of respiratory function. A Friedman's ANOVA will be used to test for differences in the EMG outcomes across the multiple (4 or more) time points. Post-hoc comparisons will be conducted using a Wilcoxon signed-rank test.
Maximal inspiratory pressure will be used to assess diaphragm strength | Change in baseline to months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  Respiratory function will be assessed using standard clinical approaches to measure inspiratory and expiratory pressures and volumes as well as standard spirometry. A Friedman's ANOVA will be used to test for differences in the respiratory outcomes across the multiple (4 or more) time points. Post-hoc comparisons will be conducted using a Wilcoxon signed-rank test.
Sniff nasal inspiratory pressure may be used to assess diaphragm strength | Change in baseline to months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  Respiratory function will be assessed using standard clinical approaches to measure inspiratory and expiratory pressures and volumes as well as standard spirometry. A Friedman's ANOVA will be used to test for differences in the respiratory outcomes across the multiple (4 or more) time points. Post-hoc comparisons will be conducted using a Wilcoxon signed-rank test.
Maximal expiratory pressure will be used to assess respiratory function | Change in baseline to months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  Respiratory function will be assessed using standard clinical approaches to measure inspiratory and expiratory pressures and volumes as well as standard spirometry. A Friedman's ANOVA will be used to test for differences in the respiratory outcomes across the multiple (4 or more) time points. Post-hoc comparisons will be conducted using a Wilcoxon signed-rank test.
Spirometry and flow volume curves/loops will be used to assess respiratory function at rest | Change in baseline to months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  Respiratory function will be assessed using standard clinical approaches to measure inspiratory and expiratory pressures and volumes as well as standard spirometry. A Friedman's ANOVA will be used to test for differences in the respiratory outcomes across the multiple (4 or more) time points. Post-hoc comparisons will be conducted using a Wilcoxon signed-rank test.
Spirometry and forced flow volume curves/loops will be used to assess respiratory function at maximal effort | Change in baseline to months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  Respiratory function will be assessed using standard clinical approaches to measure inspiratory and expiratory pressures and volumes as well as standard spirometry. A Friedman's ANOVA will be used to test for differences in the respiratory outcomes across the multiple (4 or more) time points. Post-hoc comparisons will be conducted using a Wilcoxon signed-rank test.

SECONDARY OUTCOMES:
American Spinal Cord Injury (ASIA) Impairment Scale | Change in baseline to months 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12
  Standardized clinical assessment of sensation and strength based on levels of the spinal cord to classify the severity of injury. The test is clinician-administered; clinical examination conducted to test whether sensation is 0-absent; 1-impaired or 2-normal. The lower score the worse the paralysis and the higher the score will indicate the lesser of the paralysis.

CONTACTS AND LOCATIONS:
Overall Officials: Emily J Fox, PT, DPT, PhD, Principal Investigator — University of Florida; Brooks Rehabilitation
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Brooks Rehabilitation, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Posluszny JA Jr, Onders R, Kerwin AJ, Weinstein MS, Stein DM, Knight J, Lottenberg L, Cheatham ML, Khansarinia S, Dayal S, Byers PM, Diebel L. Multicenter review of diaphragm pacing in spinal cord injury: successful not only in weaning from ventilators but also in bridging to independent respiration. J Trauma Acute Care Surg. 2014 Feb;76(2):303-9; discussion 309-10. doi: 10.1097/TA.0000000000000112. PMID 24458038
- [Background] Onders RP, Elmo M, Kaplan C, Katirji B, Schilz R. Extended use of diaphragm pacing in patients with unilateral or bilateral diaphragm dysfunction: a new therapeutic option. Surgery. 2014 Oct;156(4):776-84. doi: 10.1016/j.surg.2014.07.021. PMID 25239317
- [Background] Romero FJ, Gambarrutta C, Garcia-Forcada A, Marin MA, Diaz de la Lastra E, Paz F, Fernandez-Dorado MT, Mazaira J. Long-term evaluation of phrenic nerve pacing for respiratory failure due to high cervical spinal cord injury. Spinal Cord. 2012 Dec;50(12):895-8. doi: 10.1038/sc.2012.74. Epub 2012 Jul 10. PMID 22777487
- [Background] Hirschfeld S, Exner G, Luukkaala T, Baer GA. Mechanical ventilation or phrenic nerve stimulation for treatment of spinal cord injury-induced respiratory insufficiency. Spinal Cord. 2008 Nov;46(11):738-42. doi: 10.1038/sc.2008.43. Epub 2008 May 13. PMID 18475279
- [Background] Onders RP, Khansarinia S, Weiser T, Chin C, Hungness E, Soper N, Dehoyos A, Cole T, Ducko C. Multicenter analysis of diaphragm pacing in tetraplegics with cardiac pacemakers: positive implications for ventilator weaning in intensive care units. Surgery. 2010 Oct;148(4):893-7; discussion 897-8. doi: 10.1016/j.surg.2010.07.008. Epub 2010 Aug 24. PMID 20797750
- [Background] DiMarco AF, Onders RP, Kowalski KE, Miller ME, Ferek S, Mortimer JT. Phrenic nerve pacing in a tetraplegic patient via intramuscular diaphragm electrodes. Am J Respir Crit Care Med. 2002 Dec 15;166(12 Pt 1):1604-6. doi: 10.1164/rccm.200203-175CR. PMID 12471076